CLINICAL TRIAL: NCT03134170
Title: Impact of Adding a Pharmacist to the Health Care Team in a Federally Qualified Health Center
Brief Title: Effect of Pharmacists Treating Diabetes in a FQHC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Mary Louise Wagner, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14-805
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: pharmacist; diabetes; Preventative Care; Quality of Life
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Patients are randomized to the control or intervention group. After 12 months patients in the control group who do not have well controlled diabetes may be crossed over to the interventiobn gorup
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention): The no intervention group will serve as control group. This group will receive standard care and will be an active comparator. At the end of the study they may join the intervention group
- Intervention group (Other): The intervention group will be seen by a pharmacist iin addition to their normal provider. The pharmacist will provide medication therapy review of the patient's therapy. The pharmacist will make recommendations to make revisions in the patient's therapy.
  Interventions: Other: Pharmacist review of therapy

INTERVENTIONS:
Other: Pharmacist review of therapy — Patients who are randomized to the pharmacist group will have their treatment reviewed by a pharmacist
  Arms: Intervention group

SUMMARY:
This study is a randomized controlled cross-over trial, in the form of a proof of concept study that is designed to evaluate the health outcomes resulting from incorporating a licensed clinical pharmacist in a health care team to provide case management for diabetic patients at the Henry J Austin Health Clinic. The study uses a control group design and will feature both an experimental group and a control group. The control group, of 80 patients, will receive the standard treatment at the clinic. The experimental group, of 80 patients, will receive the standard treatment as well as Medication Therapy Management and counseling from a pharmacist. After one year the patients in the control group can cross-over to the intervention group and receive care from the pharmacist.

DETAILED DESCRIPTION:
We will put all patients into one of two groups by chance (like flipping a coin). One group of 80 patients will get the regular care at the clinic (control group). The other group of 80 patients will get their regular care at the clinic plus care by a pharmacist. The pharmacist and the regular provider will work as a team to manage the patient's drug therapy (Intervention group).

We will test the status of the patient's diabetes at each visit. Tests may include:

1. Measuring weight, heart rate, and blood pressure
2. Finger stick with a small needle to check lipid (fat) concentrations, fasting blood sugar or HbA1c
3. Examining feet, skin, and eyes
4. Reviewing the patient's diary of blood sugars, diet, and exercise history
5. Filling out a survey that measures quality of life and problems that make it hard to control your diabetes
6. Referral to other specialists such as a podiatrist (foot doctor), optometrist (eye doctor), nutritionist, and dentist

Patients will have appointments with their current provider and possibly with the pharmacist at least every 3 months. However, the total number of appointments is based on the patient's health needs. The first appointment with the pharmacist will take about one hour. Additional appointments will take about 30 minutes.

The group without the pharmacist will have regular appointment times. After 12 months in the study if the patients glucose is not well controlled they can be treated by the pharmacist for 6 months.

Final measures will be made after 12 mont

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and 74
2. Medicaid insurance
3. HbA1c of 8% or greater

Exclusion Criteria:

1. HbA1C greater than 15% because the finger stick device can not accurately read values greater than this unless the HbA1C can be confirmed with a value drawn in the laboratory.
2. Age < 18 years old or age ≥ 75 years old
3. HbA1c < 8.5% PLUS presence of one or more of the following regardless of age:

   1. Limited life expectancy
   2. History of severe hypoglycemia
4. HbA1c < 8.5% PLUS presence of one or more of the following if age ≥ 65 years old:

   1. Residency in a long-term care facility (e.g. nursing home, adult family home, etc.)
   2. ≥ 3 co-existing chronic illnesses c
   3. Impairments in ability to perform two or more instrumental activities of daily living d
   4. Mild, moderate, or severe cognitive impairment as determined by the patient's provider and Mini-Cog test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C | every 3 months for one year
  Plasma glucose control

SECONDARY OUTCOMES:
Preventative care | Baseline 6 months and 12 months
  How frequent does the patient see a dentist, podiatris, optomitrist,

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin McCarthy, PharmD, Study Chair — Rutgers, Earnest Mario School of Pharmacy
Locations (1):
- Henry J Austin Health Clinic, Trenton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
In addition, the pharacists at the clinic who are treating the have access to the patient data

REFERENCES:
- [Result] Wubben DP, Vivian EM. Effects of pharmacist outpatient interventions on adults with diabetes mellitus: a systematic review. Pharmacotherapy. 2008 Apr;28(4):421-36. doi: 10.1592/phco.28.4.421. PMID 18363526
- [Result] Wallack MC, Loafman M, Sorensen TD. The Patient Safety and Clinical Pharmacy Collaborative: improving medication use systems for the underserved. J Health Care Poor Underserved. 2012 Aug;23(3 Suppl):96-102. doi: 10.1353/hpu.2012.0143. PMID 22864490